CLINICAL TRIAL: NCT06340620
Title: Randomized Trial of Endoscopic Ultrasound Examination Using EndoSound Vision System vs. Standard Echoendoscope
Brief Title: EUS Examination Using EndoSound Vision System vs. Standard Echoendoscope
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orlando Health, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 24.017.01
Record Dates: First submitted 2024-03-15; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Disease; Pancreatic Cancer; Pancreatic Cyst; Gastrointestinal Tumor; Bile Duct Diseases; Bile Duct Cancer; Lymph Node Disease; Submucosal Tumor of Gastrointestinal Tract; Gastrointestinal Cancer
Keywords: Endoscopic ultrasound; EndoSound Vision System; Randomized trial
MeSH Terms: conditions — Pancreatic Diseases; Pancreatic Neoplasms; Pancreatic Cyst; Digestive System Neoplasms; Bile Duct Diseases; Bile Duct Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard echoendoscope (Active Comparator): Standard echoendoscope will be used and EUS examination will be performed per standard of care.
  Interventions: Device: Endoscopic ultrasound examination
- EndoSound Vision System (Active Comparator): EndoSound Vision System will be used and EUS examination will be performed per standard of care.
  Interventions: Device: Endoscopic ultrasound examination

INTERVENTIONS:
Device: Endoscopic ultrasound examination — Endoscopic ultrasound examination will be performed.

SUMMARY:
This is a randomized trial to compare the standard echoendoscope with the newly developed EndoSound Visual System in the evaluation of lesions in the gastrointestinal tract.

DETAILED DESCRIPTION:
Endoscopic ultrasound (EUS) is the gold standard for evaluation and biopsy of lesions in the pancreaticobiliary tract, subepithelial lesions in the gastrointestinal tract and luminal cancer staging due to its high sensitivity and specificity. Endoscopic ultrasound examination is performed by echoendoscopes, which are endoscopes with an ultrasound probe at the distal end to allow endoscopic ultrasound evaluation. A new endoscopic ultrasound system - the EndoSound Visual System has now been developed for endoscopic ultrasound examination. The EndoSound Visual System is a device that can be attached externally to upper gastrointestinal endoscopes, thereby converting a standard endoscope into an echoendoscope which can then be used to perform an EUS examination.

The aim of this randomized trial is to compare the standard echoendoscope with the newly developed EndoSound Visual System in the evaluation of lesions in the gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Any patient undergoing EUS examination for evaluation of the pancreas, bile duct, mediastinal or intraabdominal lymph nodes, or luminal lesions in the esophagus, stomach, duodenum or colon.

Exclusion Criteria:

* Age < 18 years.
* Unable to obtain consent for the procedure from either the patient or LAR.
* Intrauterine pregnancy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-03-25 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Rate of successful completion of the requisite EUS examination | 1 day
  Rate of successful completion of the requisite examination during EUS between the EndoSound Vision System and standard echoendoscopes will be assessed, compared as a percentage of successfully completed examinations between the standard echoendoscope and Endosound Vision System.

SECONDARY OUTCOMES:
Ease of maneuverability of the device | 1 day
  The ease of maneuverability during EUS between the EndoSound Vision System and standard echoendoscopes will be assessed, based on a rating scale of 1 to 5 (whereby 1 is the most easy to maneuver and 5 is the most difficult to maneuver).
Quality of EUS imaging | 1 day
  The quality of EUS imaging during EUS between the EndoSound Vision System and standard echoendoscopes will be assessed, based on a rating scale of 1 to 5 (whereby 1 is the best quality imaging and 5 is the worst quality imaging).
Ease of performing tissue acquisition | 1 day
  The ease of performing tissue acquisition during EUS between the EndoSound Vision System and standard echoendoscopes will be assessed, based on a rating scale of 1 to 5 (whereby 1 is the most easy to perform and 5 is the most difficult to perform).
Diagnostic adequacy of procured specimen on onsite evaluation | 7 days
  Rate of diagnostic adequacy of procured tissue specimen on onsite evaluation between the EndoSound Vision System and standard echoendoscopes.
Diagnostic adequacy of procured specimen in cell block | 7 days
  Rate of diagnostic adequacy of procured tissue specimen in cell block between the EndoSound Vision System and standard echoendoscopes.
Diagnostic accuracy of procured specimen | 7 days
  Rate of diagnostic accuracy of procured tissue specimen between the EndoSound Vision System and standard echoendoscopes.
Procedure duration | 1 day
  Duration of procedure between the EndoSound Vision System and standard echoendoscopes.
Rate of procedure-related adverse events | 7 days
  Rate of procedure-related adverse events between the EndoSound Vision System and standard echoendoscopes.
Procedure costs | 7 days
  Costs associated with the endoscopic ultrasound procedures between the EndoSound Vision System and standard echoendoscopes.

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Bang, MD MPH, Principal Investigator — Orlando Health, Digestive Health Institute
Locations (1):
- Orlando Health, Orlando, Florida, United States